CLINICAL TRIAL: NCT04700397
Title: A Validation Study of Nitroglycerin Induced Acute Drop of Pd/Pa (NTG-Pd/Pa) in Clinical Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 109-081-E
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Hypotension Symptomatic; Ischemic Heart Disease
Keywords: NTG-Pd/Pa, Fractional flow reserve, adenosine
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood sampling will perform during the FFR exam
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Repeatability group 1: The patient with systolic blood pressure above 120 mmHg, who will receive a repeatability test with 200mcg, then another 100 mcg nitroglycerine injection, with a time interval of 3 minutes apart.
  Interventions: Diagnostic Test: Nitroglycerine
- Repeatability group 2: The patient with systolic blood pressure above 120 mmHg, who will receive a repeatability test with 200mcg, then another 200 mcg nitroglycerine injection, with a time interval of 3 minutes apart.
  Interventions: Diagnostic Test: Nitroglycerine
- Repeatability group 3: The patient with systolic blood pressure above 120 mmHg, who will receive a repeatability test with 200mcg, then another 300 mcg nitroglycerine injection, with a time interval of 3 minutes apart.
  Interventions: Diagnostic Test: Nitroglycerine
- pressure-recommended doses of NTG: The patient with systolic blood pressure above 100 mmHg, who will receive the nitroglycerine injection with the dose of recommendation, adjusted according to the blood pressure.
  Interventions: Diagnostic Test: Nitroglycerine

INTERVENTIONS:
Diagnostic Test: Nitroglycerine — We aim to test the repeatability of NTG-Pd/Pa with different dosages of nitroglycerine injection.

SUMMARY:
Hyperemia with adenosine was an elemental process in FFR examination. Adenosine injection will induce some discomfort, and increase cost expenditure. Nitroglycerine will induce an acute drop of Pd/Pa, and this lowest Pd/Pa was determined as NTG-Pd/Pa. NTG-Pd/Pa has a linear relationship with FFR value and has a good diagnostic accuracy to predict FFR≤0.80 in our recent study. There is only one prospective study report on the relationship between NTG-Pd/Pa and FFR. In this study, we aim to evaluate the safety of NTG-Pd/Pa, the repeatability and dose-response of this novel index. Furthermore, we will investigate the diagnostic accuracy of NTG-Pd/Pa, with FFR≤0.8 and Resting full-cycle ratio≤0.89 as ischemic threshold respectively.

DETAILED DESCRIPTION:
Fractional flow reserve (FFR) is defined as the ratio of mean distal pressure (distal to the target lesion, Pd）to mean proximal pressure (aortic pressure, Pa) in the coronary artery(Pd/Pa) while the maximal hyperemic flow is achieved. Nowadays, FFR-guided PCI is highly recommended for the assessment of physiologic ischemia in intermediate coronary lesions. However, hyperemia with adenosine was an elemental process in FFR examination. Adenosine injection will induce some discomfort, and increase cost expenditure. Based on the clinical and physiologic outcome study, a lot of non-hyperemic indexes had been proposed, and adenosine injection could be waived. Whereas, these novel physiologic indexes are limited to the proprietary software of each vendor, curtailing clinical application. Intracoronary nitroglycerin injection was needed before each FFR assessment. Nitroglycerine will induce an acute drop of Pd/Pa, and this lowest Pd/Pa was determined as NTG-Pd/Pa. NTG-Pd/Pa has a linear relationship with FFR value and has a good diagnostic accuracy to predict FFR≤0.80 in our recent study. There is only one prospective study report on the relationship between NTG-Pd/Pa and FFR. In this study, we aim to evaluate the safety of NTG-Pd/Pa, the repeatability and dose-response of this novel index. Furthermore, we will investigate the diagnostic accuracy of NTG-Pd/Pa, with FFR≤0.8 and Resting full-cycle ratio≤0.89 as ischemic threshold respectively.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for FFR examination

Exclusion Criteria:

* Hypersensitivity to adenosine or nitroglycerine
* Severe Valvular aortic stenosis
* Resting heart rate less than 50 beats per minutes
* Systolic blood pressure less than 100 mmHg or diastolic blood pressure less than 40 mmHg
* exposure to PDE-5 inhibitors within 48 hours.
* Recent intracranial hemorrhage or brain injury

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had intermediate lesion over the coronary artery and eligible for FFR examination
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-02 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
The repeatability and dose response of NTG-Pd/Pa | 10 minutes
  Comparing the difference of NTG-Pd/Pa value after various dosage of nitroglycerine injection in the same coronary lesion

SECONDARY OUTCOMES:
Major adverse cardiac event | 2 years
  MACE including target lesion failure, target vessel failure, target vessel-related myocardial infarction, and cardiac death
Diagnostic accuracy of NTG-Pd/Pa 1 | 30 minutes
  Investigate the diagnostic accuracy of NTG-Pd/Pa, with FFR≤0.8 as ischemic threshold
Diagnostic accuracy of NTG-Pd/Pa 2 | 30 minutes
  Investigate the diagnostic accuracy of NTG-Pd/Pa, with RFR≤0.89 as ischemic threshold

OTHER OUTCOMES:
Nitroglycerine related adverse events | 1 hour
  Including symptomatic hypotension or severe headache

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Boon Jong, MD, Principal Investigator — National Taiwan University Hospital, Hsinchu Branch.
Locations (1):
- National Taiwan University Hospital Hsin-Chu branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No